CLINICAL TRIAL: NCT03144245
Title: A Phase 1, First in Human, Open Label, Dose Escalation Study of AMV564, a CD33 x CD3 Tandem Diabody in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of AMV564 in Patients With AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amphivena Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMV564-101
Record Dates: First submitted 2017-04-25; First posted 2017-05-08 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; treatment; relapsed; refractory; phase 1
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMV564 (Experimental): Continuous infusion or subcutaneous dosing of AMV564 at increasing dose levels
  Interventions: Biological: AMV564
- Combination AMV564 (Experimental): Continuous infusion or subcutaneous dosing of AMV564 at increasing dose levels in combination with pembrolizumab
  Interventions: Combination Product: AMV564 in combination with pembrolizumab

INTERVENTIONS:
Biological: AMV564 — AMV564 for administration via continuous intravenous daily infusion or subcutaneous dosing
  Arms: AMV564
Combination Product: AMV564 in combination with pembrolizumab — AMV564 for administration via continuous intravenous daily infusion or subcutaneous dosing.in combination with pembrolizumab given IV every 21 days
  Arms: Combination AMV564

SUMMARY:
This is a first in human, non randomized, open-label, dose escalation study to investigate the safety, tolerability and preliminary efficacy of AMV564.

DETAILED DESCRIPTION:
This study is a first in human, Phase 1, open label, multicenter, dose escalation study with expansion at the RP2D to evaluate the safety, tolerability and preliminary antileukemic activity of AMV564 in patients with relapsed or refractory acute myeloid leukemia (AML).

AMV564 will be given on Days 1-14 of a 4-week cycle, or Days 1-28 of a 6-week cycle,via CIV or subcutaneous administration for 1 or more treatment cycles as monotherapy or in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of signing informed consent
* Diagnosis of AML according to the World Health Organization (WHO) 2008 criteria
* Relapsed or refractory disease meeting the following criteria:

  1. Primary refractory, ie, refractory to induction with a standard intensive anthracycline/cytarabine-based regimen or a non-intensive regimen (e.g., decitabine, azacytidine, low-dose cytarabine) for patients ineligible for an intensive anthracycline/cytarabine-based therapy
  2. First untreated relapse after a first CR lasting less than 12 months or first relapse refractory to salvage therapy regardless of length of first CR; or
  3. Second or later relapse. Relapse is defined as the reappearance of leukemic blasts in the peripheral blood or ≥ 5% leukemic blasts in the bone marrow after prior achievement of a CR or CRi.

OR Patients with newly diagnosed therapy-related AML, AML progressed from antecedent MDS or CMML treated with hypomethylating agents, or de novo AML with MDS-related cytogenetic abnormalities (per 2008 WHO criteria) and who are not candidates for (or decline) intensive remission induction therapy

* No more than 3 prior induction/salvage regimens to treat active disease, and no more than 1 prior stem cell transplant. Any number of continuous cycles of therapy with an individual hypomethylating agent count as one induction or salvage regimen.
* Blasts at least 5% in bone marrow
* Peripheral white blood cell (WBC) count: no upper limit at Screening, but must be < 10 x 109/L on Day 1 prior to treatment; patients with excessive blasts may be treated with hydroxyurea to bring counts down.
* Chemistry laboratory parameters within the following range:

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x the upper limit of normal (ULN)
  2. Total bilirubin ≤ 1.5x the ULN; patients with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits.
  3. Creatinine clearance > 50 mL/min (measured or calculated by Cockcroft-Gault method)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Patients with ECOG score of 2 may be included, after discussion with the Sponsor Medical Monitor, if score is influenced by symptoms attributable to underlying AML disease.
* Willing to complete all scheduled visits and assessments at the institution administering therapy
* Able to read, understand and provide written informed consent

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

* History of, or known, central nervous system (CNS) disease involvement, or prior history of National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Grade ≥ 3 drug-related CNS toxicity
* Prior allogeneic transplant (dose escalation only)
* Prior solid organ transplantation
* Treatment with anti-thymocyte globulin (ATG) within 14 days prior to start date
* Treatment with any local or systemic antineoplastic therapy or radiation within 14 days prior to the initiation of AMV564 administration (hydroxyurea is exempted if used to reduce total WBC counts)
* Clinically significant cardiac disease,
* Pulmonary, renal, hepatic, gastrointestinal, neurological or psychiatric disease that would limit compliance with study requirements
* Evidence of active, uncontrolled, viral, bacterial, or systemic fungal infection. Prophylactic therapy according to institutional protocols is acceptable.
* Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)
* Active hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Second primary malignancy that has not been in remission for greater than 3 years. Exceptions that do not require a 3-year remission include: non-melanoma skin cancer; cervical carcinoma in situ on biopsy or squamous intraepithelial lesion on Papanicolaou (PAP) smear; localized prostate cancer (Gleason score < 6); or resected melanoma in situ.
* Major trauma or major surgery within 28 days prior to the initiation of AMV564 treatment
* Any serious underlying medical or psychiatric condition (e.g. alcohol or drug abuse), dementia or altered mental status or any issue that would impair the ability of the patient to understand informed consent or that in the opinion of the investigator would contraindicate the patient's participation in the study or confound the results of the study.
* Ability to become pregnant. However, female patients who have a negative serum or urine pregnancy test before enrollment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom; intrauterine device and condom; diaphragm with spermicidal gel and condom) during the trial and for 90 days afterward (90 days after the end of AMV564 treatment) are considered eligible.
* Male patients with partners of childbearing potential.
* Pregnant or breastfeeding women
* Is a participant or plans to participate in another interventional clinical study, while taking part in this protocol. Participation in an observational study is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Dose escalation + expansion stage: incidence of all adverse events and serious adverse events (safety and tolerability) | 42 months
  Number of participants with adverse events as a measure of safety and tolerability.
Expansion stage: Efficacy - Remission Rate | 42 months
  Proportion of participants who achieve complete remission, complete remission with incomplete recovery or partial remission

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chun, MD, Study Director — Amphivena Therapeutics, Inc.
Locations (10):
- United States (10):
  - University of California, San Francisco, San Francisco, California
  - Northwestern, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - New York Medical College, Hawthorne, New York
  - Weill Cornell Medical College, The New York Presbyterian Hospital, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, The University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No